CLINICAL TRIAL: NCT03874455
Title: Tazemetostat Expanded Access Program for Adults With Solid Tumors
Status: No longer available | Type: Expanded Access
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Other Study IDs: EZH-701
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Epithelioid Sarcoma (Ex-US Only); Spindle Cell Sarcoma; Sinonasal Carcinoma; Small Cell Carcinoma of the Ovary Hypercalcemic Type; Thoracic Sarcoma; Poorly Differentiated Chordoma; ATRT; Malignant Rhabdoid Tumor of Kidney; Malignant Rhabdoid Tumor of Ovary; Malignant Rhabdoid Tumor; Myxoid Spindle Cell Sarcoma; Epithelioid Malignant Peripheral Nerve Sheath Tumor; Chondrosarcoma; Renal Cell Carcinoma; Myoepithelial Carcinoma; Synovial Sarcoma; Renal Medullary Carcinoma; Malignant Mesothelioma; Desmoplastic Small Round Cell Tumor (DSRCT); Intramedullary Spinal Cord Schwannomatosis
MeSH Terms: conditions — Sarcoma; Rhabdoid Tumor; Chondrosarcoma; Carcinoma, Renal Cell; Sarcoma, Synovial; Mesothelioma, Malignant; Desmoplastic Small Round Cell Tumor | interventions — tazemetostat

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat (EPZ-6438) is a selective small molecule inhibitor of the histone-lysine methyltransferase EZH2 gene
  Other Names: EPZ-6438

SUMMARY:
Patients with a diagnosis listed under "conditions" below are eligible to be considered for the EAP. These conditions must be serious or life-threatening at the time of enrollment and appropriate, comparable, or satisfactory alternative treatments must have been tried without clinical success. Patients with conditions not listed under "conditions" below are not eligible for the tazemetostat EAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age (at the time of consent): >18 years of age.
2. They are unable to participate in tazemetostat clinical trials for their condition.
3. Can provide signed written informed consent.
4. Documented loss of INI1 or SMARCA4 confirmed by IHC, or molecular confirmation of tumor bi-allelic INI1 or SMARCA4 loss or mutation when INI1 or SMARCA4 IHC is equivocal or unavailable.
5. Female patients of childbearing potential should:

   * Agree to practice one highly effective method of contraception and one additional effective (barrier, for example condom or diaphragm with spermicide) method at the same time, from the time of providing voluntary written informed consent through (30 days or 5 half-lives, whichever is longer) after the last dose of tazemetostat, and
   * Have a negative beta-human chorionic gonadotropin (β-hCG) pregnancy test at time of screening and within 14 days prior to planned first dose of tazemetostat (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing), and
   * Agree to use effective contraception from start of screening until 30 days following the last dose of tazemetostat and have a male partner who uses a condom, or
   * Practice true abstinence, (when this is in line with the preferred and usual lifestyle of the patient or
   * Have a male partner who is vasectomized.
6. Male patients with a female partner of childbearing potential should:

   * Be vasectomized, or
   * Agree to use condoms from first dose of tazemetostat until 30 days following the last dose of tazemetostat, or
   * Have a female partner who is NOT of childbearing potential.

Exclusion Criteria:

1. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet and all foods that contain those fruits from time of enrollment to while on the EAP.
2. Is currently taking any prohibited medication(s) as described in section 6.3.
3. Has known hypersensitivity to any of the components of tazemetostat or other inhibitor(s) of EZH2.
4. Has thrombocytopenia, neutropenia, or anemia of grade ≥3 (per CTCAE 4.03 criteria) within the past month, or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).
5. Is known to have any abnormalities associated with MDS (e.g. del 5q, chr 7 abn) and MPN (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing.
6. Has a prior history of T-LBL/T-ALL.
7. For female patients of childbearing potential: Is pregnant or nursing.
8. For male patients: Is unwilling to adhere to contraception criteria from time of enrollment in study to at least 30 days after last dose of tazemetostat.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen